CLINICAL TRIAL: NCT00797225
Title: A Phase II, Randomized, Double-Blind, Placebo- and Active-Controlled Study to Assess the Efficacy and Safety of NBI-56418 in Subjects With Endometriosis
Brief Title: Efficacy and Safety Study of Elagolix Versus Placebo or Leuprorelin Acetate in Endometriosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-56418-0703; 2007-006474-28 (EudraCT Number)
Record Dates: First submitted 2008-11-21; First posted 2008-11-25 (Estimated); Results first posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-04

CONDITIONS: Endometriosis
Keywords: bone mineral density,endometriosis,pelvic pain
MeSH Terms: conditions — Endometriosis | interventions — elagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo tablets once a day and placebo intramuscular injection once a month for 12 weeks. At the end of 12 weeks participants were re-randomized to receive one of the two doses of elagolix (150 mg or 250 mg) for 12 weeks.
  Interventions: Drug: Placebo to Elagolix; Drug: Placebo to Leuprorelin Acetate
- Elagolix 150 mg (Experimental): Participants received elagolix 150 mg tablets once a day and placebo intramuscular injection once a month for 12 weeks. At the end of 12 weeks participants continued to receive elagolix 150 mg for an additional 12 weeks.
  Interventions: Drug: Elagolix; Drug: Placebo to Leuprorelin Acetate
- Elagolix 250 mg (Experimental): Participants received elagolix 250 mg tablets once a day and placebo intramuscular injection once a month for 12 weeks. At the end of 12 weeks participants continued to receive elagolix 250 mg for an additional 12 weeks.
  Interventions: Drug: Elagolix; Drug: Placebo to Leuprorelin Acetate
- Leuprorelin (Other): Participants received placebo tablets once a day and leuprorelin acetate 1-month depot 3.75 mg intramuscular injection once a month for 12 weeks. At the end of 12 weeks participants were re-randomized to receive one of the two doses of elagolix (150 mg or 250 mg) for 12 weeks.
  Interventions: Drug: Leuprorelin Acetate Depot; Drug: Placebo to Elagolix

INTERVENTIONS:
Drug: Leuprorelin Acetate Depot — Leuprorelin acetate depot injection 3.75 mg administered as an intramuscular injection
  Other Names: Prostap SR
  Arms: Leuprorelin
Drug: Elagolix — Elagolix tablets administered orally
  Other Names: NBI-56418; Orilissa™
  Arms: Elagolix 150 mg; Elagolix 250 mg
Drug: Placebo to Elagolix — Placebo tablet administered orally
  Arms: Leuprorelin; Placebo
Drug: Placebo to Leuprorelin Acetate — Saline solution administered as an intramuscular injection
  Arms: Elagolix 150 mg; Elagolix 250 mg; Placebo

SUMMARY:
This study is designed to evaluate the safety and beneficial effects of elagolix (NBI-56418) compared to placebo and leuprorelin (an approved endometriosis therapy) over a three month period followed by an additional three months of treatment on elagolix.

DETAILED DESCRIPTION:
The study followed a parallel-group design in which participants were randomized (1:1:1:1) to one of the following treatment groups for the first 12 weeks of dosing: 150 mg elagolix once daily (q.d.); 250 mg elagolix q.d.; placebo; or leuprorelin acetate depot injection 3.75 mg (monthly). Blinding was achieved using a double-dummy design. Following 12 weeks of dosing, participants continued in the study for an additional 12 weeks; participants randomized to elagolix continued to receive their assigned dose and participants randomized to placebo or leuprorelin acetate were re-randomized to receive one of the two doses of elagolix (150 mg q.d. or 250 mg q.d.) for 12 weeks in a double-blind fashion. Six weeks after the last dose of the study drug at the end of Week 24, a follow-up visit was performed (end of Week 30).

There was no pre-specified primary efficacy end point as there was no single key efficacy outcome measure in this exploratory Phase 2 study. For purposes of results reported here, Change From Baseline in the Monthly Mean Numerical Rating Score (NRS) for Endometriosis Pain is designated as the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria

* Female, aged 18 to 45 years, inclusive
* Have moderate to severe pelvic pain due to endometriosis
* Have been surgically (laparoscopy) diagnosed with endometriosis within the last 5 years and have recurrent or persistent endometriosis symptoms
* Have regular menstrual cycle (23-33 day)
* Agree to use two forms of non-hormonal contraception during the study

Exclusion Criteria:

* Received a Gonadotropin-releasing hormone (GnRH) agonist, GnRH antagonist, danazol, or have received any of these agents within 6 months of the start of screening.
* Received subcutaneous medroxyprogesterone acetate (DMPA-SC) or intramuscular (i.m.) medroxyprogesterone acetate (DMPA-IM), or have received either of these agents within 3 months of the start of screening.
* Are currently using hormonal contraception or other forms of hormonal therapy or received such treatment within the last month
* Have had surgery for endometriosis within the last month
* Are using systemic steroids on a chronic or regular basis within 3 months
* Have uterine fibroids or other pelvic lesions ≥ 3 cm in diameter
* Have had a hysterectomy or oophorectomy
* Have pelvic pain that is not caused by endometriosis
* Have unstable medical condition or chronic disease
* Have been pregnant within the last 6 months and is currently breast feeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2008-11-26 (Actual); Primary Completion 2010-02-24 (Actual); Study Completion 2010-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 26 November 2008 to 24 February 2010 at 27 centers in Central Eastern Europe (Bulgaria, Hungary, Poland, Romania, Russia and Ukraine).
Pre-assignment Details: Patients were randomized equally to oral elagolix 150 mg or 250 mg once daily, placebo or leuprorelin acetate (LA) 1-month depot 3.75 mg injection for 12 weeks. Thereafter, patients originally randomized to placebo or LA were re-randomized to 1 of the elagolix doses and patients randomized to elagolix continued their assigned dose for 12 weeks.
Groups:
- Placebo / Elagolix 150 mg: Participants initially randomized to placebo were re-randomized at week 12 to receive elagolix 150 mg for 12 weeks.
- Placebo / Elagolix 250 mg: Participants initially randomized to placebo were re-randomized at week 12 to receive elagolix 250 mg for 12 weeks.
- Leuprorelin / Elagolix 150 mg: Participants initially randomized to leuprorelin acetate were re-randomized at week 12 to receive elagolix 150 mg for 12 weeks.
- Leuprorelin / Elagolix 250 mg: Participants initially randomized to leuprorelin acetate were re-randomized at week 12 to receive elagolix 250 mg for 12 weeks.
Period: Weeks 1 to 12
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin | Placebo / Elagolix 150 mg | Placebo / Elagolix 250 mg | Leuprorelin / Elagolix 150 mg | Leuprorelin / Elagolix 250 mg
Started | 43 | 43 | 44 | 44 | 0 | 0 | 0 | 0
Received Study Drug | 43 | 43 | 44 | 44 | 0 | 0 | 0 | 0
Completed | 41 | 42 | 43 | 44 | 0 | 0 | 0 | 0
Not Completed | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Weeks 13 to 24
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin | Placebo / Elagolix 150 mg | Placebo / Elagolix 250 mg | Leuprorelin / Elagolix 150 mg | Leuprorelin / Elagolix 250 mg
Started | 0 | 42 | 43 | 0 | 20 | 21 | 22 | 22
Completed | 0 | 38 | 41 | 0 | 19 | 21 | 20 | 22
Not Completed | 0 | 4 | 2 | 0 | 1 | 0 | 2 | 0
Not completed — Non-compliance | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin | Total
Number analyzed (Participants) | 43 | 43 | 44 | 44 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (0.8) | 32.1 (0.9) | 31.7 (1.0) | 31.4 (0.7) | 31.7 (0.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 43 | 44 | 44 | 174
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 43 | 43 | 44 | 44 | 174

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Monthly Mean Numerical Rating Score (NRS) for Endometriosis Pain
Description: The NRS is an 11-point scale used to measure endometriosis pain and was completed at approximately the same time each day using an electronic diary (e-Diary). Participants were instructed to select a single number between 0 (No pain) and 10 (Worst pain ever) that best described their endometriosis pain at its worst over the past day.
  The monthly mean NRS is the average of the daily values reported during the 4 weeks prior to each visit.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 evaluable e-Diary report following randomization (intent-to-treat population). The analysis includes participants with non-missing data at each time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 43 | 43 | 44 | 44
units on a scale
  Week 4 | -0.35 (0.17) | -0.84 (0.17) | -1.00 (0.17) | -0.94 (0.17)
  Week 8: number analyzed (Participants) | 41 | 43 | 43 | 44
  Week 8 | -0.93 (0.20) | -1.25 (0.20) | -1.57 (0.20) | -1.55 (0.20)
  Week 12: number analyzed (Participants) | 41 | 42 | 42 | 44
  Week 12 | -1.22 (0.21) | -1.34 (0.21) | -1.47 (0.21) | -1.81 (0.20)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Analysis at Week 4. The change from baseline in monthly mean values of the NRS for overall endometriosis-associated pelvic pain was analyzed using a mixed-effects repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for participant, the baseline-by-time interaction and the baseline value as a covariate; Test type: Superiority; p = 0.0464, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.49, 95% CI 2-sided [-0.98 to -0.01], Standard Error of Mean 0.25
Statistical Analysis 2: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0080, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.65, 95% CI 2-sided [-1.13 to -0.17], Standard Error of Mean 0.24
Statistical Analysis 3: Comparison: Placebo vs Leuprorelin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0159, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.59, 95% CI 2-sided [-1.08 to -0.11], Standard Error of Mean 0.24
Statistical Analysis 4: Comparison: Placebo vs Elagolix 150 mg; Analysis at Week 8. The change from baseline in monthly mean values of the NRS for overall endometriosis-associated pelvic pain was analyzed using a mixed-effects repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for participant, the baseline-by-time interaction and the baseline value as a covariate; Test type: Superiority; p = 0.2563, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.33, 95% CI 2-sided [-0.89 to 0.24], Standard Error of Mean 0.29
Statistical Analysis 5: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.0239, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.65, 95% CI 2-sided [-1.21 to -0.09], Standard Error of Mean 0.28
Statistical Analysis 6: Comparison: Placebo vs Leuprorelin; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.0280, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.63, 95% CI 2-sided [-1.19 to -0.07], Standard Error of Mean 0.28
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg; Analysis at Week 12. The change from baseline in monthly mean values of the NRS for overall endometriosis-associated pelvic pain was analyzed using a mixed-effects repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for participant, the baseline-by-time interaction and the baseline value as a covariate; Test type: Superiority; p = 0.6904, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.12, 95% CI 2-sided [-0.70 to 0.46], Standard Error of Mean 0.29
Statistical Analysis 8: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.4022, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.25, 95% CI 2-sided [-0.83 to 0.33], Standard Error of Mean 0.29
Statistical Analysis 9: Comparison: Placebo vs Leuprorelin; [analysis description as in outcome 1, analysis 7]; Test type: Superiority; p = 0.0451, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.59, 95% CI 2-sided [-1.17 to -0.01], Standard Error of Mean 0.29

2. Secondary Outcome: Change From Baseline in the Monthly Peak Numerical Rating Score (NRS) for Endometriosis Pain
Description: The NRS is an 11-point scale used to measure endometriosis pain and was completed at approximately the same time each day using an electronic diary (e-Diary). Participants were instructed to select a single number between 0 (No pain) and 10 (Worst pain ever) that best described their endometriosis pain at its worst over the past day.
  The monthly peak NRS is the maximum of the daily values reported during the 4 weeks prior to each visit.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 43 | 43 | 44 | 44
units on a scale
  Week 4 | -0.20 (0.34) | -1.82 (0.34) | -1.83 (0.33) | -1.48 (0.33)
  Week 8: number analyzed (Participants) | 41 | 43 | 43 | 44
  Week 8 | -0.89 (0.34) | -2.23 (0.34) | -2.96 (0.33) | -3.62 (0.33)
  Week 12: number analyzed (Participants) | 41 | 42 | 42 | 44
  Week 12 | -1.67 (0.34) | -2.62 (0.34) | -3.05 (0.34) | -3.99 (0.33)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Analysis at Week 4. The change from baseline in monthly peak value of the NRS for overall endometriosis-associated pelvic pain was analyzed using a mixed-effects repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for participant, the baseline-by-time interaction and the baseline value as a covariate; Test type: Superiority; p = 0.0007, Mixed-effects Repeated Measures Model; LS Mean Difference = -1.62, 95% CI 2-sided [-2.56 to -0.69], Standard Error of Mean 0.48
Statistical Analysis 2: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0006, Mixed-effects Repeated Measures Model; LS Mean Difference = -1.63, 95% CI 2-sided [-2.56 to -0.70], Standard Error of Mean 0.47
Statistical Analysis 3: Comparison: Placebo vs Leuprorelin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0073, Mixed-effects Repeated Measures Model; LS Mean Difference = -1.28, 95% CI 2-sided [-2.21 to -0.35], Standard Error of Mean 0.47
Statistical Analysis 4: Comparison: Placebo vs Elagolix 150 mg; Analysis at Week 8. The change from baseline in monthly peak value of the NRS for overall endometriosis-associated pelvic pain was analyzed using a mixed-effects repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for participant, the baseline-by-time interaction and the baseline value as a covariate; Test type: Superiority; p = 0.0054, Mixed-effects Repeated Measures Model; LS Mean Difference = -1.34, 95% CI 2-sided [-2.28 to -0.40], Standard Error of Mean 0.48
Statistical Analysis 5: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p < 0.0001, Mixed-effects Repeated Measures Model; LS Mean Difference = -2.07, 95% CI 2-sided [-3.01 to -1.12], Standard Error of Mean 0.48
Statistical Analysis 6: Comparison: Placebo vs Leuprorelin; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p < 0.0001, Mixed-effects Repeated Measures Model; LS Mean Difference = -2.73, 95% CI 2-sided [-3.67 to -1.79], Standard Error of Mean 0.48
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg; Analysis at Week 12. The change from baseline in monthly peak value of the NRS for overall endometriosis-associated pelvic pain was analyzed using a mixed-effects repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for participant, the baseline-by-time interaction and the baseline value as a covariate; Test type: Superiority; p = 0.0509, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.95, 95% CI 2-sided [-1.89 to 0.00], Standard Error of Mean 0.48
Statistical Analysis 8: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; p = 0.0046, Mixed-effects Repeated Measures Model; LS mean Difference = -1.38, 95% CI 2-sided [-2.33 to -0.43], Standard Error of Mean 0.48
Statistical Analysis 9: Comparison: Placebo vs Leuprorelin; [analysis description as in outcome 2, analysis 7]; Test type: Superiority; p < 0.0001, Mixed-effects Repeated Measures Model; LS Mean Difference = -2.32, 95% CI 2-sided [-3.26 to -1.38], Standard Error of Mean 0.48

3. Secondary Outcome: Change From Baseline in the Monthly Mean Non-menstrual Pelvic Pain Score
Description: Participants assessed their pelvic pain not related to menses and its impact on their daily activities at approximately the same time every day in an e-Diary according to the following response options:
  * 0 = No pelvic pain
  * 1 = Mild pelvic pain; subject could not do some of the things she usually does
  * 2 = Moderate pelvic pain; subject could not do many of the things she usually does
  * 3 = Severe pelvic pain; subject could not do most or all of the things she usually does.
  The monthly mean non-menstrual pelvic pain score is the average of the daily values reported during the 4 weeks prior to each visit.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 43 | 43 | 44 | 44
units on a scale
  Week 4 | -0.05 (0.06) | -0.22 (0.06) | -0.21 (0.06) | -0.27 (0.06)
  Week 8: number analyzed (Participants) | 41 | 43 | 43 | 44
  Week 8 | -0.18 (0.06) | -0.34 (0.06) | -0.36 (0.06) | -0.46 (0.06)
  Week 12: number analyzed (Participants) | 41 | 42 | 42 | 44
  Week 12 | -0.30 (0.06) | -0.35 (0.06) | -0.34 (0.06) | -0.55 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Analysis at Week 4. The change from baseline in monthly mean non-menstrual pelvic pain scores was analyzed using a mixed-effects repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for participant, the baseline-by-time interaction and the baseline value as a covariate; Test type: Superiority; p = 0.0453, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.16, 95% CI 2-sided [-0.33 to 0.00], Standard Error of Mean 0.08
Statistical Analysis 2: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0609, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.15, 95% CI 2-sided [-0.31 to 0.01], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Placebo vs Leuprorelin; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0069, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.22, 95% CI 2-sided [-0.38 to -0.06], Standard Error of Mean 0.08
Statistical Analysis 4: Comparison: Placebo vs Elagolix 150 mg; Analysis at Week 8. The change from baseline in monthly mean non-menstrual pelvic pain scores was analyzed using a mixed-effects repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for participant, the baseline-by-time interaction and the baseline value as a covariate; Test type: Superiority; p = 0.0556, Mixed-effects Repeated Measures Model]; LS Mean Difference = -0.16, 95% CI 2-sided [-0.32 to 0.00], Standard Error of Mean 0.08
Statistical Analysis 5: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.0387, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.17, 95% CI 2-sided [-0.33 to -0.01], Standard Error of Mean 0.08
Statistical Analysis 6: Comparison: Placebo vs Leuprorelin; [analysis description as in outcome 3, analysis 4]; Test type: Superiority; p = 0.0008, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.28, 95% CI 2-sided [-0.44 to -0.12], Standard Error of Mean 0.08
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg; Analysis at Week 12. The change from baseline in monthly mean non-menstrual pelvic pain scores was analyzed using a mixed-effects repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for participant, the baseline-by-time interaction and the baseline value as a covariate; Test type: Superiority; p = 0.5879, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.04, 95% CI 2-sided [-0.21 to 0.12], Standard Error of Mean 0.08
Statistical Analysis 8: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.6122, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.04, 95% CI 2-sided [-0.20 to 0.12], Standard Error of Mean 0.08
Statistical Analysis 9: Comparison: Placebo vs Leuprorelin; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.0023, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.25, 95% CI 2-sided [-0.41 to -0.09], Standard Error of Mean 0.08

4. Secondary Outcome: Change From Baseline in the Monthly Mean Dysmenorrhea Score
Description: Participants assessed dysmenorrhea (pain during menstruation) and its impact on their daily activities at approximately the same time each day of their period in an e-Diary according to the following response options:
  * Subject is not having her period
  * 0 = No pain related to period
  * 1 = Mild pain related to period; subject could not do some of the things she usually does
  * 2 = Moderate pain related to period; subject could not do many of the things she usually does
  * 3 = Severe pain related to period; subject could not do most of or all of the things she usually does.
  The monthly mean dysmenorrhea score is the average of the daily values reported during the 4 weeks prior to each visit.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 43 | 43 | 44 | 44
units on a scale
  Week 4 | -0.17 (0.08) | -0.64 (0.08) | -0.67 (0.08) | -0.65 (0.08)
  Week 8: number analyzed (Participants) | 41 | 43 | 43 | 44
  Week 8 | -0.40 (0.08) | -0.86 (0.08) | -1.04 (0.08) | -1.22 (0.08)
  Week 12: number analyzed (Participants) | 41 | 42 | 42 | 44
  Week 12 | -0.35 (0.08) | -0.76 (0.08) | -0.87 (0.08) | -1.14 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Analysis at Week 4. The change from baseline in monthly mean dysmenorrhea scores was analyzed using a mixed-effects repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for participant, the baseline-by-time interaction and the baseline value as a covariate; Test type: Superiority; p < 0.0001, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.47, 95% CI 2-sided [-0.69 to -0.24], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Mixed-effects Repeated Measures Model; LS mean Difference = -0.50, 95% CI 2-sided [-0.73 to -0.27], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Placebo vs Leuprorelin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.48, 95% CI 2-sided [-0.71 to -0.25], Standard Error of Mean 0.12
Statistical Analysis 4: Comparison: Placebo vs Elagolix 150 mg; Analysis at Week 8. The change from baseline in monthly mean dysmenorrhea scores was analyzed using a mixed-effects repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for participant, the baseline-by-time interaction and the baseline value as a covariate; Test type: Superiority; p < 0.0001, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.46, 95% CI 2-sided [-0.69 to -0.23], Standard Error of Mean 0.12
Statistical Analysis 5: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 4, analysis 4]; Test type: Superiority; p < 0.0001, Mixed-effects Repeated Measures Model; LS mean Difference = -0.64, 95% CI 2-sided [-0.87 to -0.40], Standard Error of Mean 0.12
Statistical Analysis 6: Comparison: Placebo vs Leuprorelin; [analysis description as in outcome 4, analysis 4]; Test type: Superiority; p < 0.0001, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.82, 95% CI 2-sided [-1.04 to -0.59], Standard Error of Mean 0.12
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg; Analysis at Week 12. The change from baseline in monthly mean dysmenorrhea scores was analyzed using a mixed-effects repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for participant, the baseline-by-time interaction and the baseline value as a covariate; Test type: Superiority; p = 0.0005, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.41, 95% CI 2-sided [-0.65 to -0.18], Standard Error of Mean 0.12
Statistical Analysis 8: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 4, analysis 7]; Test type: Superiority; p < 0.0001, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.52, 95% CI 2-sided [-0.76 to -0.29], Standard Error of Mean 0.12
Statistical Analysis 9: Comparison: Placebo vs Leuprorelin; [analysis description as in outcome 4, analysis 7]; Test type: Superiority; p < 0.0001, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.79, 95% CI 2-sided [-1.02 to -0.56], Standard Error of Mean 0.12

5. Secondary Outcome: Change From Baseline in the Monthly Mean Sum of Dysmenorrhea and Non-menstrual Pelvic Pain Scores
Description: Participants assessed dysmenorrhea and pelvic pain not related to menses and their impact on daily activities at approximately the same time every day on a 4-point scale (0 = none, 1 = mild, 2 = moderate, and 3 = severe) in an e-Diary. The dysmenorrhea scale included an option for participants who were not having their period.
  The sum of the dysmenorrhea and non-menstrual pelvic pain scores on each day were calculated to create a daily total score. On days the participant was not having her period, the dysmenorrhea score was not defined; hence, the total score was equal to the non-menstrual pelvic pain score (range 0 to 3). On days where the participant recorded menstruation the total score ranged from 0 to 6, where higher scores indicate more severe pain. The monthly mean sum of dysmenorrhea and non-menstrual pelvic pain scores is the average of the daily values reported during the 4 weeks prior to each visit.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 43 | 43 | 44 | 44
units on a scale
  Week 4 | -0.12 (0.07) | -0.43 (0.07) | -0.44 (0.07) | -0.50 (0.07)
  Week 8: number analyzed (Participants) | 41 | 43 | 43 | 44
  Week 8 | -0.24 (0.07) | -0.58 (0.07) | -0.67 (0.07) | -0.78 (0.07)
  Week 12: number analyzed (Participants) | 41 | 42 | 42 | 44
  Week 12 | -0.40 (0.07) | -0.55 (0.07) | -0.63 (0.07) | -0.87 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Elagolix 150 mg; Analysis at Week 4. The change from baseline in monthly mean sum of dysmenorrhea and non-menstrual pelvic pain scores was analyzed using a mixed-effects repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for participant, the baseline-by-time interaction and the baseline value as a covariate; Test type: Superiority; p = 0.0011, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.32, 95% CI 2-sided [-0.51 to -0.13], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0010, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.32, 95% CI 2-sided [-0.51 to -0.13], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: Placebo vs Leuprorelin; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.38, 95% CI 2-sided [-0.57 to -0.19], Standard Error of Mean 0.10
Statistical Analysis 4: Comparison: Placebo vs Elagolix 150 mg; Analysis at Week 8. The change from baseline in monthly mean sum of dysmenorrhea and non-menstrual pelvic pain scores was analyzed using a mixed-effects repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for participant, the baseline-by-time interaction and the baseline value as a covariate; Test type: Superiority; p = 0.0007, Mixed-effects Repeated Measures Model; -0.33 = -0.33, 95% CI 2-sided [-0.52 to -0.14], Standard Error of Mean 0.10
Statistical Analysis 5: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p < 0.0001, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.43, 95% CI 2-sided [-0.62 to -0.24], Standard Error of Mean 0.10
Statistical Analysis 6: Comparison: Placebo vs Leuprorelin; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p < 0.0001, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.54, 95% CI 2-sided [-0.73 to -0.35], Standard Error of Mean 0.10
Statistical Analysis 7: Comparison: Placebo vs Elagolix 150 mg; Analysis at Week 12. The change from baseline in monthly mean sum of dysmenorrhea and non-menstrual pelvic pain scores was analyzed using a mixed-effects repeated measures analysis of covariance model. The model included fixed effects for treatment, time, the treatment-by-time interaction, a random effect for participant, the baseline-by-time interaction and the baseline value as a covariate; Test type: Superiority; p = 0.1319, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.15, 95% CI 2-sided [-0.34 to 0.04], Standard Error of Mean 0.10
Statistical Analysis 8: Comparison: Placebo vs Elagolix 250 mg; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.0222, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.22, 95% CI 2-sided [-0.42 to -0.03], Standard Error of Mean 0.10
Statistical Analysis 9: Comparison: Placebo vs Leuprorelin; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p < 0.0001, Mixed-effects Repeated Measures Model; LS Mean Difference = -0.47, 95% CI 2-sided [-0.66 to -0.28], Standard Error of Mean 0.10

6. Secondary Outcome: Change From Baseline in the Percentage of Days of Any Analgesic Use
Description: The daily use of endometriosis analgesics was reported by participants daily using the e-Diary. Participants reported whether the medication was over-the-counter (OTC) or prescription, and, if prescription, whether the medication was a narcotic.
  The percentage of days of any analgesic use is defined as the number of days in the 4 weeks prior to each study visit that the participant reported the use of an analgesic, divided by the number of study days in the interval that the participant provided an e-Diary report regarding the use of endometriosis analgesics (including a response of "none").
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 43 | 43 | 44 | 44
percentage of days
  Week 4 | -5.2 (2.0) | -1.1 (2.0) | -8.4 (2.0) | -8.7 (2.0)
  Week 8: number analyzed (Participants) | 41 | 43 | 43 | 44
  Week 8 | -6.2 (2.0) | -3.4 (2.0) | -9.1 (2.0) | -10.2 (2.0)
  Week 12: number analyzed (Participants) | 41 | 42 | 42 | 44
  Week 12 | -6.2 (2.0) | -4.4 (2.0) | -8.3 (2.0) | -10.5 (2.0)

7. Secondary Outcome: Change From Baseline in the Percentage of Days of Prescription Analgesic Use
Description: The daily use of endometriosis analgesics was reported by participants daily using the e-Diary. Participants reported whether the medication was over-the-counter (OTC) or prescription, and, if prescription, whether the medication was a narcotic.
  The percentage of days of prescription analgesic use is defined as the number of days in the 4 weeks prior to each study visit that the participant reported the use of a prescription analgesic, divided by the number of study days in the interval that the participant provided an e-Diary report regarding the use of endometriosis analgesics (including a response of "none").
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 43 | 43 | 44 | 44
percentage of days
  Week 4 | -0.3 (1.8) | 3.4 (1.8) | -1.2 (1.7) | -2.5 (1.7)
  Week 8: number analyzed (Participants) | 41 | 43 | 43 | 44
  Week 8 | -1.3 (1.6) | 1.3 (1.6) | -2.8 (1.6) | -2.6 (1.6)
  Week 12: number analyzed (Participants) | 41 | 42 | 42 | 44
  Week 12 | -1.8 (1.4) | 0.7 (1.4) | -1.9 (1.4) | -2.8 (1.3)

8. Secondary Outcome: Change From Baseline in the Percentage of Days of Narcotic Analgesic Use
Description: The daily use of endometriosis analgesics was reported by participants daily using the e-Diary. Participants reported whether the medication was over-the-counter (OTC) or prescription, and, if prescription, whether the medication was a narcotic.
  The percentage of days of narcotic analgesic use is defined as the number of days in the 4 weeks prior to each study visit that the participant reported the use of a narcotic analgesic, divided by the number of study days in the interval that the participant provided an e-Diary report regarding the use of endometriosis analgesics (including a response of "none").
Time Frame: Baseline, Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 43 | 43 | 44 | 44
percentage of days
  Week 4 | 0.0 (0.1) | -0.1 (0.1) | 0.0 (0.1) | -0.1 (0.1)
  Week 8: number analyzed (Participants) | 41 | 43 | 43 | 44
  Week 8 | -0.1 (0.1) | -0.1 (0.1) | -0.1 (0.1) | -0.1 (0.1)
  Week 12: number analyzed (Participants) | 41 | 42 | 42 | 44
  Week 12 | 0.0 (0.1) | 0.1 (0.1) | 0.1 (0.1) | 0.3 (0.1)

9. Secondary Outcome: Change From Baseline in Dyspareunia Component of the Composite Pelvic Signs and Symptoms Score (CPSSS)
Description: The CPSSS consists of 5 components that address dysmenorrhea, dyspareunia, non-menstrual pelvic pain, pelvic tenderness, and pelvic induration.
  To assess dyspareunia (painful intercourse) participants were asked to select the best description of pain during sexual intercourse over the past 28 days using the following response categories:
  * 0 = Absent; No discomfort during sexual intercourse.
  * 1 = Mild; I can tolerate the discomfort during sexual intercourse.
  * 2 = Moderate; Intercourse is sometime interrupted due to pain.
  * 3 = Severe; I prefer to avoid intercourse because of pain.
  * Not applicable. I am not sexually active for reasons other than my endometriosis symptoms.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 evaluable e-Diary report following randomization (intent-to-treat population). The analysis includes participants with non-missing data at baseline and at each time point.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 40 | 38 | 40 | 41
units on a scale
  Week 4: number analyzed (Participants) | 38 | 36 | 39 | 39
  Week 4 | -0.33 (0.11) | -0.46 (0.11) | -0.49 (0.11) | -0.55 (0.11)
  Week 8: number analyzed (Participants) | 37 | 36 | 39 | 38
  Week 8 | -0.72 (0.11) | -0.68 (0.11) | -0.77 (0.11) | -0.76 (0.11)
  Week 12: number analyzed (Participants) | 37 | 33 | 40 | 37
  Week 12 | -0.60 (0.11) | -0.84 (0.12) | -0.89 (0.11) | -1.04 (0.11)

10. Secondary Outcome: Change From Baseline in Dysmenorrhea Component of the CPSSS
Description: The CPSSS consists of 5 components that address dysmenorrhea, dyspareunia, non-menstrual pelvic pain, pelvic tenderness, and pelvic induration.
  To assess dysmenorrhea (pain during menstruation), participants were asked to select the best description of painful menstruation over the past 28 days using the following response categories:
  * 0 = Absent; Amenorrhea (no bleeding) or no discomfort.
  * 1 = Mild; Some loss of work efficiency; occasional use of analgesics.
  * 2 = Moderate; In bed part of one day, occasional loss of work; regular use of analgesics.
  * 3 = Severe; In bed ≥ 1 day, incapacitation; requirement for strong analgesics.
Time Frame: Baseline and Week 12
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 evaluable e-Diary report following randomization (intent-to-treat population). Data collection for this endpoint was added via a protocol amendment; therefore, the analysis only includes the subset of participants affected by the protocol amendment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 20 | 19 | 23 | 24
units on a scale | -1.03 (0.17) | -1.29 (0.17) | -1.47 (0.16) | -1.75 (0.15)

11. Secondary Outcome: Change From Baseline in Non-menstrual Pelvic Pain CPSSS Component
Description: The CPSSS consists of 5 components that address dysmenorrhea, dyspareunia, non-menstrual pelvic pain, pelvic tenderness, and pelvic induration.
  To assess non-menstrual pelvic pain, participants were asked to select the best description of pelvic pain over the past 28 days using the following response categories:
  * 0 = Absent; No discomfort.
  * 1 = Mild; Occasional pelvic discomfort that can be treated with NSAIDs.
  * 2 = Moderate; Noticeable discomfort or pain for most of cycle requiring regular use of NSAID or weak opiate.
  * 3 = Severe; Pain persisting during the cycle or pain requiring strong analgesics.
Time Frame: Baseline and Week 12
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 20 | 19 | 23 | 24
units on a scale | -0.60 (0.12) | -0.58 (0.12) | -0.48 (0.11) | -0.79 (0.11)

12. Secondary Outcome: Patient Global Impression of Change at Weeks 4, 8 and 12
Description: The Patient Global Impression of Change (PGIC) is a questionnaire-based assessment of the change in endometriosis pain since the initiation of study drug. The participant was asked to select from one of seven response categories:
  1. Very Much Improved
  2. Much Improved
  3. Minimally Improved
  4. Not Changed
  5. Minimally Worse
  6. Much Worse
  7. Very Much Worse
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 43 | 43 | 44 | 44
units on a scale
  Week 4: number analyzed (Participants) | 41 | 43 | 43 | 44
  Week 4 | 3.4 (0.1) | 3.0 (0.1) | 2.9 (0.2) | 3.3 (0.1)
  Week 8: number analyzed (Participants) | 41 | 43 | 43 | 44
  Week 8 | 2.8 (0.1) | 2.5 (0.2) | 2.2 (0.1) | 2.3 (0.1)
  Week 12: number analyzed (Participants) | 41 | 42 | 43 | 44
  Week 12 | 2.6 (0.2) | 2.4 (0.1) | 2.2 (0.2) | 2.1 (0.1)

13. Secondary Outcome: Percentage of Participants With a PGIC Response of Minimally Improved, Much Improved, or Very Much Improved
Description: The PGIC is a questionnaire-based assessment of the change in endometriosis pain since the initiation of study drug. The participant was asked to select from one of seven response categories:
  1. Very Much Improved
  2. Much Improved
  3. Minimally Improved
  4. Not Changed
  5. Minimally Worse
  6. Much Worse
  7. Very Much Worse
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 43 | 43 | 44 | 44
percentage of participants
  Week 4: number analyzed (Participants) | 41 | 43 | 43 | 44
  Week 4 | 56.1 [40.9 to 71.3] | 74.4 [61.4 to 87.5] | 65.1 [50.9 to 79.4] | 50.0 [35.2 to 64.8]
  Week 8: number analyzed (Participants) | 41 | 43 | 43 | 44
  Week 8 | 75.6 [62.5 to 88.8] | 81.4 [69.8 to 93.0] | 90.7 [82.0 to 99.4] | 88.6 [79.3 to 98.0]
  Week 12: number analyzed (Participants) | 41 | 42 | 43 | 44
  Week 12 | 80.5 [68.4 to 92.6] | 88.1 [78.3 to 97.9] | 88.4 [78.8 to 98.0] | 93.2 [85.7 to 100.0]

14. Secondary Outcome: Percentage of Participants With a PGIC Response of Much Improved or Very Much Improved
Description: as for outcome 13
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 43 | 43 | 44 | 44
percentage of participants
  Week 4: number analyzed (Participants) | 41 | 43 | 43 | 44
  Week 4 | 7.3 [0.0 to 15.3] | 25.6 [12.5 to 38.6] | 32.6 [18.6 to 46.6] | 27.3 [14.1 to 40.4]
  Week 8: number analyzed (Participants) | 41 | 43 | 43 | 44
  Week 8 | 36.6 [21.8 to 51.3] | 53.5 [38.6 to 68.4] | 72.1 [58.7 to 85.5] | 54.5 [39.8 to 69.3]
  Week 12: number analyzed (Participants) | 41 | 42 | 43 | 44
  Week 12 | 53.7 [38.4 to 68.9] | 54.8 [39.7 to 69.8] | 67.4 [53.4 to 81.4] | 70.5 [57.0 to 83.9]

15. Secondary Outcome: Change From Baseline in Endometriosis Health Profile-5 (EHP-5) at Week 12
Description: The EHP-5 is an instrument to measure health-related quality of life in women with endometriosis. The EHP-5 consists of two parts:
  * A core questionnaire consisting of five questions that measure the areas of pain, control and powerlessness, emotional well-being, social support, and self-image with five response categories for each item (Never, Rarely, Sometimes, Often, Always)
  * A supplemental questionnaire consisting of six additional questions which assess the areas of work, relationship with children, sexual intercourse, feelings about the medical profession, treatment, and infertility with the same five response categories plus an additional response category of Not Relevant which was not scored.
  The scores associated with each possible outcome category are as follows: never (0), rarely (25), sometimes (50), often (75), and always (100). A negative change from baseline score indicates improvement in quality of life.
Time Frame: Baseline and week 12
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 evaluable e-Diary report following randomization (intent-to-treat population). The analysis includes participants with non-missing data for each dimension at baseline and week 12.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 43 | 43 | 44 | 44
units on a scale
  Pain: number analyzed (Participants) | 41 | 42 | 43 | 44
  Pain | -14.0 (4.8) | -19.0 (4.1) | -25.0 (4.7) | -31.8 (3.9)
  Control and Powerlessness: number analyzed (Participants) | 41 | 42 | 43 | 44
  Control and Powerlessness | -18.3 (4.4) | -17.9 (3.9) | -20.9 (5.1) | -23.9 (4.9)
  Emotional Wellbeing: number analyzed (Participants) | 41 | 42 | 43 | 44
  Emotional Wellbeing | -14.6 (4.2) | -10.7 (4.1) | -12.8 (4.4) | -13.6 (4.4)
  Social Support: number analyzed (Participants) | 41 | 42 | 43 | 44
  Social Support | -22.0 (4.4) | -16.1 (4.4) | -18.6 (5.6) | -15.3 (5.1)
  Self-image: number analyzed (Participants) | 41 | 42 | 43 | 44
  Self-image | -12.2 (6.5) | -7.7 (4.5) | -5.8 (5.0) | -8.5 (4.1)
  Work: number analyzed (Participants) | 39 | 36 | 36 | 35
  Work | -23.7 (3.9) | -21.5 (4.5) | -29.9 (5.1) | -38.6 (4.3)
  Relationship with Children: number analyzed (Participants) | 13 | 18 | 16 | 12
  Relationship with Children | -11.5 (6.7) | -15.3 (5.4) | -25.0 (7.6) | -22.9 (9.5)
  Sexual Intercourse: number analyzed (Participants) | 38 | 33 | 40 | 38
  Sexual Intercourse | -32.2 (5.7) | -21.2 (6.2) | -30.6 (5.3) | -28.9 (5.7)
  Medical Profession: number analyzed (Participants) | 33 | 32 | 33 | 32
  Medical Profession | -5.3 (4.5) | -5.5 (4.0) | -7.6 (3.0) | -6.3 (4.2)
  Frustration with Treatment: number analyzed (Participants) | 22 | 23 | 23 | 22
  Frustration with Treatment | -11.4 (6.1) | -10.9 (6.3) | -7.6 (6.9) | -12.5 (6.9)
  Concerns with Infertility: number analyzed (Participants) | 33 | 25 | 29 | 30
  Concerns with Infertility | -19.7 (5.0) | -24.0 (7.0) | -13.8 (5.2) | -13.3 (4.8)

16. Secondary Outcome: Concentration of Serum Estradiol
Description: The concentration of serum estradiol (E2) was quantified using liquid chromatography with tandem mass spectrophotometry (LC/MS/MS). Serum estradiol concentrations below the limit of quantification (BLQ) were set equal to the lower limit of quantification (2.5 pg/mL).
Time Frame: Baseline and Weeks 4, 8 and 12
Population: Randomized participants who received at least one dose of randomized, double-blind study drug with at least one eDiary value following randomization, excluding participants who had less than 80% oral study drug dosing compliance during Weeks 1-12 (per protocol population). The analysis includes participants with non-missing data at each time point.
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 43 | 41 | 43 | 44
pg/mL
  Baseline: number analyzed (Participants) | 43 | 41 | 43 | 43
  Baseline | 39.10 [12.0 to 168.0] | 43.40 [2.5 to 199.0] | 47.50 [12.4 to 497.0] | 46.20 [19.6 to 154.0]
  Week 4: number analyzed (Participants) | 42 | 40 | 43 | 42
  Week 4 | 49.50 [14.6 to 436.0] | 36.40 [4.5 to 247.0] | 22.00 [6.2 to 127.0] | 3.63 [2.5 to 87.5]
  Week 8: number analyzed (Participants) | 41 | 39 | 42 | 42
  Week 8 | 61.00 [12.7 to 440.0] | 36.90 [6.8 to 182.0] | 23.65 [2.5 to 213.0] | 4.36 [2.5 to 44.9]
  Week 12: number analyzed (Participants) | 27 | 41 | 41 | 30
  Week 12 | 87.90 [2.5 to 338.0] | 36.70 [2.5 to 521.0] | 26.20 [2.5 to 235.0] | 6.38 [2.5 to 421.0]

17. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Femur at Week 12
Description: Bone mineral density (BMD) of the femur (total hip) was measured by dual-energy X-ray absorptiometry (DXA).
Time Frame: Baseline and week 12
Population: Participants who received at least one dose of randomized, double-blind study drug (safety analysis set) and with available BMD data at baseline and week 12.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 40 | 41 | 42 | 43
percent change | -0.90 (1.316) | -0.342 (1.583) | -0.5623 (1.367) | -1.122 (1.634)

18. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Spine at Week 12
Description: Bone mineral density (BMD) of the spine was measured by dual-energy X-ray absorptiometry (DXA).
Time Frame: Baseline and week 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 40 | 41 | 42 | 44
percent change | 0.106 (1.893) | -1.053 (1.985) | -0.799 (2.352) | -1.633 (2.113)

19. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Femur at Week 24
Description: Bone mineral density (BMD) of the femur (total hip) was measured by dual-energy X-ray absorptiometry (DXA).
Time Frame: Baseline and Week 24
Population: Participants who received at least one dose of randomized, double-blind study drug (safety analysis set) and with available BMD data at baseline and week 24.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Elagolix 150 mg | Elagolix 250 mg | Placebo / Elagolix 150 mg | Placebo / Elagolix 250 mg | Leuprorelin / Elagolix 150 mg | Leuprorelin / Elagolix 250 mg
Number analyzed (Participants) | 36 | 38 | 17 | 20 | 18 | 21
percent change | -0.549 (1.827) | -0.699 (1.574) | -0.126 (1.732) | -0.573 (1.328) | -1.784 (1.571) | -1.783 (2.096)

20. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density of the Spine at Week 24
Description: Bone mineral density (BMD) of the spine was measured by dual-energy X-ray absorptiometry (DXA).
Time Frame: Baseline and Week 24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Elagolix 150 mg | Elagolix 250 mg | Placebo / Elagolix 150 mg | Placebo / Elagolix 250 mg | Leuprorelin / Elagolix 150 mg | Leuprorelin / Elagolix 250 mg
Number analyzed (Participants) | 35 | 39 | 17 | 20 | 18 | 21
percent change | -1.288 (2.681) | -1.855 (2.670) | -0.990 (2.636) | -0.648 (2.377) | -2.899 (2.733) | -4.378 (2.099)

21. Secondary Outcome: Change From Baseline in Serum N-telopeptide Concentration at Week 12
Description: Blood samples to determine N-telopeptide concentrations were analyzed by a central laboratory using an enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline and week 12
Population: Participants who received at least one dose of randomized, double-blind study drug (safety analysis set) and with available data at baseline and week 12.
Measure: Mean (Standard Error); unit: nM bone collagen equivalents (BCE)
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 39 | 43 | 41 | 40
nM bone collagen equivalents (BCE) | 0.62 (0.78) | 0.77 (0.69) | 2.04 (0.66) | 3.18 (0.72)

22. Secondary Outcome: Average Number of Hot Flashes Per Day
Description: Hot flashes, if any, were reported daily by participants during the study using the e-Diary.
  The average number of hot flashes per day was calculated for each participant as the total number of hot flashes divided by total days in the phase.
Time Frame: Screening (8 weeks prior to day 1), Treatment phase (weeks 1 to 12 for participants in the placebo and leuprorelin treatment groups and weeks 1 to 24 for participants in the elagolix treatment groups)
Population: Participants who received at least one dose of randomized, double-blind study drug (safety analysis set).
Measure: Median (Full Range); unit: hot flashes per day
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 43 | 43 | 44 | 44
hot flashes per day
  Screening | 0.00 [0.0 to 4.8] | 0.00 [0.0 to 4.6] | 0.00 [0.0 to 2.6] | 0.00 [0.0 to 3.7]
  Treatment Phase | 0.11 [0.0 to 3.0] | 0.22 [0.0 to 7.5] | 1.10 [0.0 to 11.4] | 1.73 [0.0 to 9.4]

23. Secondary Outcome: Percentage of Days With Uterine Bleeding
Description: Uterine bleeding was reported daily by participants during the study using the e-Diary.
  The percentage of days a participant reported any bleeding was calculated as the total number of days the participant reported any bleeding ( light, moderate, or heavy) divided by the total number of days the participant had a non-missing eDiary report of vaginal bleeding in the phase.
Time Frame: as for outcome 22
Population: Participants who received at least one dose of randomized, double-blind study drug (safety analysis set).
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin
Number analyzed (Participants) | 43 | 43 | 44 | 44
percentage of days
  Screening | 21.10 (1.78) | 18.32 (1.14) | 22.32 (1.68) | 21.05 (1.87)
  Treatment Phase | 21.46 (1.39) | 10.78 (1.14) | 9.54 (1.35) | 11.04 (1.30)

24. Secondary Outcome: Number of Days to First Posttreatment Menses
Description: Defined as the number of days from the last dose of study drug until the start date of the first post-treatment menses.
Time Frame: From last day of study drug up to 6 weeks after the last dose.
Population: Participants who received at least one dose of randomized, double-blind study drug (safety analysis set) with non-missing post-treatment data.
Measure: Median (Full Range); unit: days
Arm/Group | Elagolix 150 mg | Elagolix 250 mg | Placebo / Elagolix 150 mg | Placebo / Elagolix 250 mg | Leuprorelin / Elagolix 150 mg | Leuprorelin / Elagolix 250 mg
Number analyzed (Participants) | 38 | 39 | 19 | 20 | 20 | 21
days | 22.5 [3 to 56] | 26.0 [10 to 103] | 26.0 [5 to 42] | 27.0 [2 to 34] | 29.0 [5 to 62] | 28.0 [8 to 36]

ADVERSE EVENTS:
Time Frame: From the first dose of any study drug through week 30. The Placebo and Leuprorelin treatment groups include data for the initial 12-week treatment phase. The Elagolix treatment groups include data for the 24 week treatment period plus 6 weeks follow-up for participants initially randomized to elagolix, and 12 week treatment period plus 6-week follow-up for participants initially randomized to placebo or leuprorelin and were re-randomized at week 12.
Groups:
- Placebo: Participants received placebo tablets once a day and placebo intramuscular injection once a month for 12 weeks.
- Elagolix 150 mg: Participants initially randomized to elagolix 150 mg received elagolix 150 mg tablets once a day and placebo intramuscular injection once a month for 12 weeks. At the end of 12 weeks participants continued to receive elagolix 150 mg for an additional 12 weeks.
  Participants initially randomized to placebo or leuprorelin were re-randomized at week 12 to receive elagolix 150 mg for 12 weeks.
- Elagolix 250 mg: Participants initially randomized to elagolix 250 mg received elagolix 250 mg tablets once a day and placebo intramuscular injection once a month for 12 weeks. At the end of 12 weeks participants continued to receive elagolix 250 mg for an additional 12 weeks.
  Participants initially randomized to placebo or leuprorelin were re-randomized at week 12 to receive elagolix 250 mg for 12 weeks.
- Leuprorelin Acetate: Participants received placebo tablets once a day and leuprorelin acetate 1-month depot 3.75 mg intramuscular injection once a month for 12 weeks.
Arm/Group | Placebo | Elagolix 150 mg | Elagolix 250 mg | Leuprorelin Acetate
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/85 | 0/87 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/43 | 1/85 | 2/87 | 0/44
Other Adverse Events (participants affected / at risk) | 3/43 | 25/85 | 21/87 | 6/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=43) | Elagolix 150 mg (N=85) | Elagolix 250 mg (N=87) | Leuprorelin Acetate (N=44)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIABETES MELLITUS NON-INSULIN-DEPENDENT (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PARANASAL SINUS BENIGN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=43) | Elagolix 150 mg (N=85) | Elagolix 250 mg (N=87) | Leuprorelin Acetate (N=44)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 6 (6) | 2 (2) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 6 (6) | 5 (5) | 0 (0)
BONE DENSITY DECREASED (Investigations) | 0 (0) | 7 (7) | 6 (6) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (2) | 11 (21) | 10 (12) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.